CLINICAL TRIAL: NCT00001363
Title: Functional Brain Mapping of Planning Activities With [015] Water PET Blood Flow Technique
Brief Title: PET Scan to Map the Areas of the Brain Involved in Planning
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930077; 93-N-0077
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Cognition Disorders
Keywords: Blood Flow; Chess Play; Frontal Lobe; Neurobehavioral Deficits; Neuropsychology; Positron Emission Tomography; Prefrontal Cortex
MeSH Terms: conditions — Cognition Disorders

SUMMARY:
Positron Emission Tomography (PET) is a technique used to investigate the functional activity of the brain. The PET technique allows doctors to study the normal processes of the brain (central nervous system) of normal individuals and patients with neurologic illnesses without physical / structural damage to the brain.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases blood flow to and from the area of activity increases also. Knowing these facts, researchers can use radioactive water (H215O) and PET scans to observe what areas of the brain are receiving more blood flow.

This study will attempt to determine the areas of the brain activated by planning processes and decision making. Researchers will ask patients to participate in tests and games (chess) that will stimulate the areas of the brain involved with decision making and planning while undergoing the water PET blood flow technique.

DETAILED DESCRIPTION:
This protocol will attempt to determine the topographical distribution in the brain of the cognitive components of planning using the [150] water PET blood flow technique. We will administer perception, motor, simple decision, and planning tasks using the game of chess and the Tower of Hanoi Test as paradigms. Utilizing a "subtraction technique" we hope to identify those areas of cerebral cortex which are most activated by planning processes. It is predicted that the dorsolateral frontal areas will be most prominently activated. It is also predicted that the essential components of the planning process will be the same regardless of the type of plans being executed. The data we collect will be of value in determining 1) the neural representation of planning processes and 2) in guiding cognitive models of the planning system.

ELIGIBILITY:
Normal Controls:

Males and female subjects from two age ranges: 18-30 and 50-65 years of age.

Individuals with a history of neurological or psychiatric disorder will not be included nor will individuals currently taking psychoactive medication.

Patients:

Patients with outstanding problems in planning.

Patients must have a diagnosed CNS disorder with lesion localization verified by MRI scanning available from the referring physician or completed at the NIH Clinical Center.

Patients with unilateral or bilateral lesions that meet the behavioral criteria for selection (planning disorder).

Patients will be medication free (or taking medication with no known central nervous system effects) and be able to understand instructions and task demands.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230
Dates: Start 1993-01; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Nichelli P, Grafman J, Pietrini P, Alway D, Carton JC, Miletich R. Brain activity in chess playing. Nature. 1994 May 19;369(6477):191. doi: 10.1038/369191a0. No abstract available. PMID 8183339
- [Background] Partiot A, Grafman J, Sadato N, Flitman S, Wild K. Brain activation during script event processing. Neuroreport. 1996 Feb 29;7(3):761-6. doi: 10.1097/00001756-199602290-00020. PMID 8733740
- [Background] Flitman S, O'Grady J, Cooper V, Grafman J. PET imaging of maze processing. Neuropsychologia. 1997 Apr;35(4):409-20. doi: 10.1016/s0028-3932(96)00086-3. PMID 9106270